CLINICAL TRIAL: NCT01835197
Title: A Phase 1, Within Cohort, Randomized, Double Blind, Third-Party Open, Placebo-Controlled, Single- And Multiple Dose Escalation, Parallel Group Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-04965842 In Healthy Western and Japanese Subjects
Brief Title: First-in-Human Study to Evaluate Safety and Tolerability of Single and Multiple Ascending Doses of Janus Kinase-1 Inhibitor PF-04965842 in Healthy Western and Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7451001
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Phase 1; Randomized; Double Blind; Placebo-Controlled; Single- & Multiple Dose Escalation; Safety; Tolerability; PK; PD; Pf-04965842
MeSH Terms: interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- SAD Cohorts 1-8 Experimental Arm (Experimental)
  Interventions: Drug: PF-04965842
- SAD Cohorts 1-8 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- MAD Cohorts 3 through 5 Experimental Arm (Experimental)
  Interventions: Drug: PF-04965842
- MAD Cohorts 3 through 5 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- MAD Cohorts 6 and 7 Experimental Arm (Experimental)
  Interventions: Drug: PF-04965842
- MAD Cohorts 6 and 7 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- MAD Cohort 8 Experimental Arm (Experimental)
  Interventions: Drug: PF-04965842
- MAD Cohort 8 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- MAD Cohort 9 Experimental Arm (Experimental)
  Interventions: Drug: PF-04965842
- MAD Cohort 9 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04965842 — Subjects will receive single doses of 3, 10, 30, 100, 200, 400, or 800 mg of PF-04695842 (solution or suspension) in a dose escalation format.
  Arms: SAD Cohorts 1-8 Experimental Arm
Drug: Placebo — Subjects will receive single doses of PF-04695842 matching placebo (solution or suspension) in a dose escalation format.
  Arms: SAD Cohorts 1-8 Placebo Arm
Drug: PF-04965842 — Subjects will receive doses of 30, 100 or 200 mg (solution or suspension) once daily for 10 days.
  Arms: MAD Cohorts 3 through 5 Experimental Arm
Drug: Placebo — Subjects will receive PF-04965842 matching placebo (solution or suspension) once daily for 10 days.
  Arms: MAD Cohorts 3 through 5 Placebo Arm
Drug: PF-04965842 — Subjects will receive doses of 100 or 200 mg (suspension or solution) twice daily for 10 days.
  Arms: MAD Cohorts 6 and 7 Experimental Arm
Drug: Placebo — Subjects will receive PF-04965842 matching placebo doses (suspension or solution) twice daily for 10 days.
  Arms: MAD Cohorts 6 and 7 Placebo Arm
Drug: PF-04965842 — Subjects will receive 200 mg dose (suspension or solution) twice daily for 10 days.
  Arms: MAD Cohort 8 Experimental Arm
Drug: Placebo — Subjects will receive PF-04965842 matching placebo dose (suspension or solution) twice daily for 10 days.
  Arms: MAD Cohort 8 Placebo Arm
Drug: PF-04965842 — Subjects will receive 400 mg dose (suspension or solution) once daily for 10 days.
  Arms: MAD Cohort 9 Experimental Arm
Drug: Placebo — Subjects will receive PF-04965842 matching placebo dose (suspension or solution) once daily for 10 days.
  Arms: MAD Cohort 9 Placebo Arm

SUMMARY:
This single- and multiple-ascending dose study is the first evaluation of PF-04965842, a Janus kinase1 (JAK1) inhibitor, in humans. The goal is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics in healthy Western and Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.
* Females must be of non-child bearing potential and either at least 1 year post menopausal (FSH ≥40 IU/L), or have documented hysterectomy (with or without bilateral oophrectomy) at least 6 months prior to study day
* Subjects willing to defer receiving prophylactic immunizations (e.g. influenza or pneumococcal vaccines) during the study.
* Absolute lymphocyte count must be greater than or equal to the lower limit of the laboratory reference range.
* Subjects enrolled in Cohort 8 must have four Japanese grandparents born in Japan.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, , pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* History of hepatitis or positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBc Ab) or hepatitis C antibodies (HCV).
* Clinically significant abnormality on chest X-ray performed at screening or within 3 months of screening date; or history of tuberculosis or active or latent or inadequately treated infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline vital signs (blood pressure, pulse rate, oral temperature and respiration rate) and physical examinations | 6 weeks
Changes from baseline in 12 lead ECG parameters | 6 weeks
  Quantitative changes in ECG intervals
Incidence and severity of treatment emergent adverse events and withdrawals due to treatment emergent adverse events | 6 weeks
Incidence and magnitude of treatment emergent clinical laboratory abnormalities including hematology (with white blood cell count differentials, platelets, PT and aPTT), chemistry, fasting glucose, urinalysis | 6 weeks
Change from baseline in immunoglobulin levels | 6 weeks
  Quantitative IgG, IgA, IgM, and IgE levels
24-hour urine creatinine clearance (Single Ascending Dose Period) | Baseline, Day 1
24-hour urine creatinine clearance (Multiple Ascending Dose Period) | Baseline, Day 1

SECONDARY OUTCOMES:
Complement Level: C3 | 6 weeks
Complement Level: C4 | 6 weeks
Complement Level: C3A | 6 weeks
  Cohorts 1-7 and Cohort 9
Complement Level: Bb | 6 weeks
  Cohorts 1-7 and Cohort 9
Single Ascending Dose: Dose-normalized Area Under the Curve From Time Zero to Infinity (AUCinf(dn)) | 8 days
Multiple Ascending Dose: Accumulation Ratio based on Cmax (Rac(Cmax)) | 6 weeks
Urinary Pharmacokinetics; for twice-a-day dosing, amount of PF-0496842 excreted unchanged in 12 hours (AE12) | 6 weeks
Urinary Pharmacokinetics; for twice-a-day dosing, percent of PF-0496842 excreted unchanged in 12 hours (AE12%) | 6 weeks
Multiple Ascending Dose: Apparent Volume of Distribution at Steady State (Vz/F) | 6 weeks
  Vz/F is the distribution of a drug between plasma and the rest of the body following oral adminstration.
Multiple Ascending Dose: Apparent Total Body Clearance (CL/F) | 6 weeks
Urinary Pharmacokinetics; for once-a-day dosing, amount of PF-0496842 excreted unchanged in 24 hours (AE24) | 6 weeks
Urinary Pharmacokinetics; for once-a-day dosing, percent of PF-0496842 excreted unchanged in 24 hours (AE24%) | 6 weeks
Renal Clearance (CLr) | 6 weeks
High-Sensitivity C-Reactive Protein (hsCRP) | 6 weeks
Neutrophil counts | 6 weeks
Reticulocyte counts | 6 weeks
Complement Level: CH50 | 6 weeks
Single Ascending Dose: Apparent Total Body Clearance (CL/F) | 8 days
Multiple Ascending Dose: Maximum Observed Plasma Concentration (Cmax) | 6 weeks
Multiple Ascending Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax) | 6 weeks
Multiple Ascending Dose: Dose-normalized Maximum Observed Plasma Concentration (Cmax(dn)) | 6 weeks
Multiple Ascending Dose: Area Under the Curve to the end of the dosing period (AUCtau(dn)) | 6 weeks
Multiple Ascending Dose: Accumulation Ratio based on AUC predicted (Rss) | 6 weeks
Multiple Ascending Dose: Accumulation Ration based on AUC observed (Rac) | 6 weeks
Multiple Ascending Dose: Plasma Decay Half-Life (t1/2) | 6 weeks
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one-half.
Multiple Ascending Dose: Peak to Trough Fluctuation (PTF) | 6 weeks
Single Ascending Dose: Dose-normalized Area Under the Curve to the end of the dosing period (AUCtau(dn)) | 8 days
Single Ascending Dose: Area Under the Curve From Time Zero to Infinity (AUCinf) | 8 days
Single Ascending Dose: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 8 days
Single Ascending Dose: Dose-normalized Maximum Observed Plasma Concentration (Cmax(dn)) | 8 days
Single Ascending Dose: Area Under the Curve to the end of the dosing period (AUCtau) | 8 days
Single Ascending Dose: Dose-normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast(dn)) | 8 days
  Dose-normalized area under the plasma concentration time-curve from zero to the last measured concentration (AUClast(dn))
Single Ascending Dose: Plasma Decay Half-Life (t1/2) | 8 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Multiple Ascending Dose: Area Under the Curve to the end of the dosing period (AUCtau) | 6 weeks
Single Ascending Dose: Apparent Volume of Distribution (Vz/F) | 8 days
Single Ascending Dose: Maximum Observed Plasma Concentration (Cmax) | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- [Derived] Peeva E, Hodge MR, Kieras E, Vazquez ML, Goteti K, Tarabar SG, Alvey CW, Banfield C. Evaluation of a Janus kinase 1 inhibitor, PF-04965842, in healthy subjects: A phase 1, randomized, placebo-controlled, dose-escalation study. Br J Clin Pharmacol. 2018 Aug;84(8):1776-1788. doi: 10.1111/bcp.13612. Epub 2018 May 24. PMID 29672897
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7451001&StudyName=First-in-Human%20Study%20to%20Evaluate%20Safety%20and%20Tolerability%20of%20Single%20and%20Multiple%20Ascending%20Doses%20of%20Janus%20Kinase-1%20Inhibitor%20PF-04965842%20in